CLINICAL TRIAL: NCT03750084
Title: Anaesthesia and mHealth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Annelies De Cock, Data nurse, Universitair Ziekenhuis Brussel
Other Study IDs: ANESmHealth
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia; Cell Phone; Mobile Applications
Keywords: Anesthesia; Cell Phone; Mobile Applications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionary — The intervention consists of a digitally distributed questionary.

SUMMARY:
This survey aims to better define the wishes/needs of the Belgian Anaesthesiologists within the field of mobile technology, namely, what would help improve the daily anaesthesia practice.

DETAILED DESCRIPTION:
This study consists of a simple online survey that takes approximately 3 minutes to complete.

The study aims to assess the confidence of the belgian anaesthesiologists on smartphone applications and dedicated smartphone peripherals, on how these can be used in daily practice, as well as what their wishes for further developments are.

ELIGIBILITY:
Inclusion Criteria:

* Active diploma-holding Anesthesiologist working in Belgium

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Active diploma-holding Anesthesiologists working in Belgium
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire about the Confidence (scale 0-5) on Mobile Apps and Peripheral Devices in Anesthesiology | One single time-point assessment (time of filling in the questionnaire) during 3 months (time during which the filling-in of the questionnaire is possible)
  Confidence of Anesthesiologist on the use of Mobile Apps and Peripheral Devices in improving anesthesia care.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Carvalho, MD, MSc, Principal Investigator — Universitair Ziekenhuis Brussel; Jan Poelaert, MD, PhD, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
No intention to share.

REFERENCES:
- [Derived] Carvalho H, Verdonck M, Forget P, Poelaert J. Acceptance of mHealth among health professionals: a case study on anesthesia practitioners. BMC Anesthesiol. 2020 Mar 3;20(1):55. doi: 10.1186/s12871-020-00958-3. PMID 32126985